CLINICAL TRIAL: NCT05482802
Title: The Exploration of an Active Training Tool to Reduce Weight Bias Among Students Pursuing a Healthcare-related Degree
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Principal investigator, Ariel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU-HEA-SSD-20220709
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Obesity Bias
MeSH Terms: conditions — Weight Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An active training tool on weight bias and knowledge about obesity (Active Comparator): The intervention will take place at the university simulation center and include three components. First, a short-lecture on obesity and weight bias. Second, four scenarios that simulate meetings between health professionals and people with obesity which will be presented by professional role-players in sequence. Each scenario will include a different therapeutic situation and include varying degrees of weight bias, stigma, and discrimination to stimulate students to think and react. Third, an active open discourse with a person with obesity will be held.
  Interventions: Behavioral: An active training tool on weight bias and knowledge about obesity
- A short-written document on obesity (Placebo Comparator): A short-written document on obesity which will be based on current literature.
  Interventions: Behavioral: A short-written document on obesity

INTERVENTIONS:
Behavioral: An active training tool on weight bias and knowledge about obesity — The intervention will take place at the university simulation center and include three components. First, a short lecture on obesity and weight bias. Second, four scenarios that simulate meetings between health professionals and people with obesity which will be presented by professional role-players in sequence. Each scenario will include a different therapeutic situation and include varying degrees of weight bias, stigma, and discrimination to stimulate students to think and react. Third, an active open discourse with a person with obesity will be held.
  Arms: An active training tool on weight bias and knowledge about obesity
Behavioral: A short-written document on obesity — A short-written document on obesity which will be based on current literature.
  Arms: A short-written document on obesity

SUMMARY:
An open-label parallel RCT will be conducted among 220 students pursuing a health-related degree at Ariel university. The intervention tool will be based on the constructive social learning model and will include a short lecture on obesity, scenarios simulating a meeting between health professionals and patients with obesity that will be presented by professional role-players and include varying degrees of weight bias, stigma and discrimination, and an open discourse with a patient with obesity. The tool's development will be carried out throughout recommended steps including a comprehensive literature review, preparation of a preliminary draft of the plan, evaluation of the planned intervention tool in terms of content validity, and a pilot testing of the tool among n=15 students from the target population.

The control group will receive a short-written document on obesity. This study will utilize an embedded mixed-method approach. At baseline, one- and six- weeks post-intervention both groups will be asked to fill an anonymous online survey which will include demographics, weight and body perception, knowledge about obesity, the Anti-Fat Attitudes questionnaire, the Short-Form of Fat-Phobia scale, and the Weight-Implicit Association-Test. Moreover, in-depth interviews will be conducted among 15 participants from each group.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students pursuing a healthcare-related degree including nutrition science, health systems management, communication disorders, physiotherapy, occupational therapy, and nursing at Ariel university
* age ≥18 years
* willingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Anti-Fat Attitudes questionnaire ('AFA') | Change from baseline at six- weeks post-intervention
  The 'AFA' indicates explicit anti-fat attitudes toward people with obesity and is composed of 13-items rated on a 10-point Likert scale and divided into three subscales ('dislike', 'fear about fat' and 'willpower'), with higher total scores indicating stronger anti-fat attitudes.
The short-form of fat-phobia scale (' F-scale') | Change from baseline at six- weeks post-intervention
  The 'F-scale' indicates fat-phobic attitudes toward people with obesity and is composed of 14-pairs of adjectives that are used to describe people with obesity (e.g., 'no willpower' vs. 'has willpower') and ranked on a 1-5 scale according to the point closest to the adjective name that describes their feelings and beliefs. Higher scores indicate stronger fat-phobic attitudes.
Weight Implicit Association Test ('IAT') | Change from baseline at six- weeks post-intervention
  IAT tool is an indirect measure of implicit bias toward weight which uses the constructs of "fat people" versus "thin people" and the polarized attitudes of "good" and "bad" to detect implicit weight bias.

SECONDARY OUTCOMES:
Knowledge about obesity | Change from baseline at six- weeks post-intervention
  Knowledge about obesity will be assessed by five questions that were written by the research team according to current literature.

OTHER OUTCOMES:
Demographics | At baseline
  Questions regarding age, gender, occupation, marital status, religious affiliation, department of studies.
Body perception | At baseline
  Body Appreciation Scale-2 is a 10-item scale which ranked on a 1-5 scale and assesses acceptance and/or favorable opinions towards a person's body.
Weight perception | At baseline
  Questions regarding self-definition of weight status, the importance of weight to self-confidence, and much control a person has over the weight.
Weight history | At baseline
  Questions regarding current weight and height, obesity during childhood, obesity during last decade, family members who struggle with obesity, currently in any process of losing weight.
Objective weight measurement | At baseline
  Measurement of actual weight in kilograms.
Objective height measurement | At baseline
  Measurement of actual height in meters.
Semi structured interviews | At six- weeks post-intervention
  Fifteen participants from each study group will be randomly chosen for conducting a semi-structured interviews. The interviews will take place six weeks post-intervention and will provide in-depth, detailed information regarding the participants' views of obesity and stigma after conducting the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shiri Sherf-Dagan, PhD, Principal Investigator — Ariel university and Assuta medical center
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sherf-Dagan S, Ofri L, Tayar I, Keisar I, Buch A, Paska-Davis N, Pinus M, Tesler R, Elran-Barak R, Boaz M, Green G. A multifaceted training tool to reduce weight bias among healthcare students: A randomized controlled trial. Obes Res Clin Pract. 2024 Jan-Feb;18(1):35-42. doi: 10.1016/j.orcp.2023.12.002. Epub 2024 Jan 5. PMID 38184475